CLINICAL TRIAL: NCT01525433
Title: Cervical Cancer Screening and Adherence to Follow-up Among Hispanic Women
Brief Title: Cervical Cancer Screening Among Hispanic Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FHCRC IR 7290; U54CA153502 (NIH)
Record Dates: First submitted 2012-01-31; First posted 2012-02-03 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention)
- Low Intensity Information (DVD) (Active Comparator): A low-intensity information program, consisting of a video approach educating women on the importance of cervical cancer screening;
  Interventions: Behavioral: DVD
- High Intensity Information (Promotora) (Active Comparator): A higher intensity information program consisting of the video plus a 'promotora' or lay-community health educator led-intervention at the participant's home to encourage cervical cancer screening.
  Interventions: Behavioral: Promotora

INTERVENTIONS:
Behavioral: DVD — Participants will received a mailed DVD containing culturally appropriate information about the importance of cervical cancer screening
  Arms: Low Intensity Information (DVD)
Behavioral: Promotora — Participants will receive a home visit from a lay community health educator ('Promotora') and will be shown a DVD containing culturally appropriate information to educate participants about the importance of cervical cancer screening
  Arms: High Intensity Information (Promotora)

SUMMARY:
In this study, 400 Hispanic women will be recruited and randomized to one of three interventions:

1. Control (no change);
2. A low-intensity information program, consisting of a video approach educating women on the importance of cervical cancer screening;
3. A higher intensity program consisting of the video plus a 'promotora' or lay-community health educator led intervention at the participant's home to encourage cervical cancer screening.

The investigators will compare which intervention is most effective in encouraging Hispanic women to undergo cervical cancer screening (Pap test)

ELIGIBILITY:
Inclusion Criteria:

* Female
* 21 - 64 years of age
* Hispanic or Latina
* Resident of the Yakima Valley, WA, USA
* No hysterectomy
* Last PAP test (cervical screening) more than 3 years ago
* Last seen at the local clinic less than 5 years ago

Exclusion Criteria:

* Less than 21 or greater than 64 years of age
* PAP test less 3 years ago
* Prior hysterectomy

Ages: 21 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 451 (Actual)
Dates: Start 2011-09; Primary Completion 2015-09 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Participant attends cervical cancer screening | Within 7 months of the intervention

SECONDARY OUTCOMES:
Patient Navigator | Elapsed time from diagnosis to clinic visit
  Evaluation of the patient navigator program as a method to improve adherence and reduce time to follow-up among study participants who receive an abnormal Pap test result. Time to follow-up will be compared to a similar population of patients who were not part of the study who also receive a diagnosis of an abnormal Pap test.

CONTACTS AND LOCATIONS:
Overall Officials: Beti Thompson, PhD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Duggan C, Coronado G, Martinez J, Byrd TL, Carosso E, Lopez C, Benavides M, Thompson B. Cervical cancer screening and adherence to follow-up among Hispanic women study protocol: a randomized controlled trial to increase the uptake of cervical cancer screening in Hispanic women. BMC Cancer. 2012 May 6;12:170. doi: 10.1186/1471-2407-12-170. PMID 22559251